CLINICAL TRIAL: NCT05069870
Title: A Three-part, Single-center, Open-label, Phase I Drug-drug Interaction Clinical Study to Investigate the Effect of Itraconazole, Gemfibrozil or Rifampicin on Pharmacokinetics of SKLB1028 in Healthy Subjects
Brief Title: A Study to Investigate the Drug-drug Interactions (DDIs) of SKLB1028 With Itraconazole, Gemfibrozil or Rifampicin in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HA114-CSP-009
Record Dates: First submitted 2021-09-15; First posted 2021-10-06 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — SKLB1028; Itraconazole; Gemfibrozil; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The DDI of SKLB1028 and Itraconazole (Experimental): Eligible subjects received a single dose of SKLB1028 100 mg on Day 1, then took Itraconazole 200 mg twice-daily on Day 8 and 200 mg once-daily on Day 9 through Day 18, and took a single dose of SKLB1028 100 mg on Day 11.
  Interventions: Drug: SKLB1028; Drug: Itraconazole
- The DDI of SKLB1028 and Gemfibrozil (Experimental): Eligible subjects received a single dose of SKLB1028 100 mg on Day 1, then took Gemfibrozil 600 mg twice-daily on Day 8 through Day 19, and took a single dose of SKLB1028 100 mg on Day 12.
  Interventions: Drug: SKLB1028; Drug: Gemfibrozil
- The DDI of SKLB1028 and Rifampicin (Experimental): Eligible subjects received a single dose of SKLB1028 150 mg on Day 1, then took Rifampicin 600 mg once-daily on Day 8 through Day22, and took a single dose of SKLB1028 150 mg on Day 15.
  Interventions: Drug: SKLB1028; Drug: Rifampicin

INTERVENTIONS:
Drug: SKLB1028 — SKLB1028, capsule, oral
Drug: Itraconazole — Itraconazole, capsule, oral
  Arms: The DDI of SKLB1028 and Itraconazole
Drug: Gemfibrozil — Gemfibrozil, capsule, oral
  Arms: The DDI of SKLB1028 and Gemfibrozil
Drug: Rifampicin — Rifampicin, capsule, oral
  Arms: The DDI of SKLB1028 and Rifampicin

SUMMARY:
This is a three-part, single-center, open-label phase I clinical study to characterize the DDIs potential of SKLB1028 with Itraconazole, Gemfibrozil or Rifampicin in healthy subjects. This study also aims to evaluate the safety and tolerability of SKLB1028 in the presence of Itraconazole, Gemfibrozil or Rifampicin.

DETAILED DESCRIPTION:
SKLB1028 is the potential substrate of CYP3A4, CYP2C8 and P-gp. This study conducted in three parts to characterize the DDIs potential of SKLB1028 with the perpetrator drugs ( Itraconazole, Gemfibrozil, Rifampicin) in Healthy Subjects. Each part of this study consists of a screening period (Day -14 to Day -2), a baseline period (Day -1), a treatment period, and a follow-up visit period.

ELIGIBILITY:
Inclusion Criteria:

-

Healthy subjects:

1. Voluntarily sign the informed consent form, understand the trial procedures, and be willing to comply with all trial procedures and restrictions;
2. 18 ≤ age ≤45, male;
3. Subjects with weight ≥50.0 kg and body mass index (BMI) 19-26 kg/m^2 (inclusive);
4. Subjects are willing to use effective contraceptives and not allowed to donate sperm from screening to the 6 months after the last dose administration unless permanent contraception has been taken, such as vasectomy.
5. Ability to communicate well with researchers, and be willing to comply with all trial requirements.

Exclusion Criteria:

1. Allergic constitution, including a history of allergy to any of the study drugs or other similarly structured drugs;
2. Previous or current severe diseases, such as cardiovascular, respiratory, gastrointestinal, endocrine, hematological, psychiatric/neurological systems diseases, or any other disease that can interfere with the results of the study;
3. Subjects who have previously undergone surgery that may affect the absorption, distribution, metabolism, or excretion of the drug (e.g., subtotal gastrectomy), or who have a scheduled surgical plan during the study period;
4. Use of any strong inhibitors or inducers of CYP3A4, CYP2C8 or P-gp within 2 weeks prior to screening;
5. Use of any prescription drug, over-the-counter drug, herbal medicine or health products within 2 weeks prior to screening;
6. History of drug abuse within 1 year prior to screening, or positive urine drug screen at screening;
7. Smoking more than 5 cigarettes per day within 6 months prior to screening;
8. Average daily intake of alcohol more than 14 units (14 units ≈285 mL of beer, or 25 mL of liquor, or 150 mL of wine) within 4 weeks prior to screening, or a positive ethanol breath test at screening;
9. Consumption of grapefruit juice, methylxanthine-rich food or beverage (such as coffee, tea, cola, chocolate, energy drinks) within 48 h before the administration, or those who have had strenuous exercise, or have other factors affecting absorption, distribution, metabolism, excretion, etc of the drug;
10. Participation in another clinical trial within 3 months before screening (whichever is administrated);
11. Blood donation (or blood loss) ≥200 mL within 4 weeks prior to the screening, or who have a blood donation plan during the entire study or within 1 months after the study;
12. Any abnormalities of clinical significance in physical examination, vital signs, clinical laboratory tests (routine blood test, blood biochemistry, routine urine test, coagulation function), anteroposterior chest radiograph or chest CT scan;
13. Abnormalities of clinical significance in 12-lead ECG examination (such as tachycardia/bradycardia in need of medical treatment, II-III degree atrioventricular block, QTcF>450 ms or any other clinically significant abnormalities );
14. Any positive test result of hepatitis B surface antigen or hepatitis C virus antibody, or subjects with a history of hepatitis B;
15. Any positive test result of anti-human immunodeficiency virus antibody or anti-Treponema pallidum specific antibody;
16. Any condition that, in the opinion of the Investigator, may prevent the subject from completing the study or poses a significant risk to the subject.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) of SKLB1028 | Up to 22 days
Area under the concentration-time curve (AUC) from 0 to the last measurable concentration (AUC0-t) of SKLB1028 | Up to 22 days
AUC extrapolated to infinity (AUCinf) of SKLB1028 | Up to 22 days

SECONDARY OUTCOMES:
Time to Cmax (Tmax) of SKLB1028 | Up to 22 days
Terminal elimination half-life (t1/2) of SKLB1028 | Up to 22 days
Apparent Clearance (CLz/F) of SKLB1028 | Up to 22 days
Apparent volume of distribution (Vz/F) of SKLB1028 | Up to 22 days
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Up to approximately 30 days
Clinically significant changes from baseline in routine blood test were recorded as AEs at each visit time point. | Up to approximately 30 days
  Routine blood test included cell count (white blood cells, platelets, basophils, eosinophils, neutrophils, lymphocytes and monocytes) in 10^9/L.
Clinically significant changes from baseline in routine blood test were recorded as AEs at each visit time point. | Up to approximately 30 days
  Routine blood test included red blood cell count in 10^12/L.
Clinically significant changes from baseline in routine blood test were recorded as AEs at each visit time point. | Up to approximately 30 days
  Routine blood test included hemoglobin in g/L.
Clinically significant changes from baseline in blood biochemistry test were recorded as AEs at each visit time point. | Up to approximately 30 days
  Blood biochemistry test included total bilirubin and serum creatinine in μmol/L.
Clinically significant changes from baseline in blood biochemistry test were recorded as AEs at each visit time point. | Up to approximately 30 days
  Blood biochemistry test included alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase and creatine kinase in U/L.
Clinically significant changes from baseline in blood biochemistry test were recorded as AEs at each visit time point. | Up to approximately 30 days
  Blood biochemistry test included total protein and albumin in g/L.
Clinically significant changes from baseline in blood biochemistry test were recorded as AEs at each visit time point. | Up to approximately 30 days
  Blood biochemistry test included total cholesterol, triglyceride and blood glucose in mmol/L.
Clinically significant changes from baseline in routine urine test were recorded as AEs at each visit time point. | Up to approximately 30 days
  Routine urine test included protein, urobilinogen, glucose and ketones (positive or negative).
Clinically significant changes from baseline in routine urine test were recorded as AEs at each visit time point. | Up to approximately 30 days
  Routine urine test included pH value and specific gravity.
Clinically significant changes from baseline in coagulation function test were recorded as AEs at each visit time point. | Up to approximately 30 days
  Coagulation function test included prothrombin time and activated partial thromboplastin time in seconds.
Clinically significant changes from baseline in coagulation function test were recorded as AEs at each visit time point. | Up to approximately 30 days
  Coagulation function test included antithrombin III as percentage.
Clinically significant changes from baseline in coagulation function test were recorded as AEs at each visit time point. | Up to approximately 30 days
  Coagulation function test included fibrinogen in g/L.
Clinically significant changes from baseline in 12-lead electrocardiogram (ECG) examination were recorded as AEs at each visit time point. | Up to approximately 30 days
  ECG monitoring included heart rate in bpm.
Clinically significant changes from baseline in 12-lead electrocardiogram (ECG) examination were recorded as AEs at each visit time point. | Up to approximately 30 days
  ECG monitoring included P-R, QRS, QT and QTcF in ms.
Clinically significant changes from baseline in vital signs examination were recorded as AEs at each visit time point. | Up to approximately 30 days
  Vital signs monitoring included body temperature in degrees Celsius.
Clinically significant changes from baseline in vital signs examination were recorded as AEs at each visit time point. | Up to approximately 30 days
  Vital signs monitoring included respiratory rate and pulse in times per minute.
Clinically significant changes from baseline in vital signs examination were recorded as AEs at each visit time point. | Up to approximately 30 days
  Vital signs monitoring included systolic blood pressure and diastolic blood pressure in mmHg.
Clinically significant changes from baseline in physical examination were recorded as AEs at each visit time point. | Up to approximately 30 days
  Physical examination included general conditions, skin, mucous membranes, head, neck, chest, abdomen, spine, limbs, nervous system, and lymphatic system.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, China